CLINICAL TRIAL: NCT06245135
Title: Short-term Effects of a Virtual, Community-based, Task-oriented Group Exercise Program Compared to a Waitlist Control in Increasing Function Among Adults With Balance and Mobility Limitations: The TIME™ at Home Randomized Controlled Trial
Brief Title: TIME™ at Home Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other); March of Dimes, Canada (Other); Heart and Stroke Foundation of Canada (Other); University of Alberta (Other); University of Manitoba (Other); Bruyère Health Research Institute. (Other)
Responsible Party: Principal Investigator, Dr. Nancy Salbach, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 45343
Record Dates: First submitted 2024-01-29; First posted 2024-02-07 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Mobility Limitation
Keywords: Virtual Exercise; Community-based Exercise; Mobility; Balance; Randomized Controlled Trial
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Outcomes Assessor
Masking Description: Single: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIME at Home (Experimental): TIME at Home is a virtual, group, task-oriented exercise program targeting balance and mobility. A community organization delivers two 1.5-hour sessions per week, for 8 weeks using Zoom.
  Interventions: Behavioral: TIME at Home
- Waitlist (No Intervention): Individuals in the waitlist control group will receive the TIME at Home program following the final 5-month evaluation.

INTERVENTIONS:
Behavioral: TIME at Home — Sessions involve a 15-minute pre-video safety check and social time; streaming a 1-hour pre-recorded exercise video; and a 15-minute post-video social time. Two trained facilitators run each class, with a maximum group size of 10 people.
  The 1-hour exercise videos include a seated warm-up and cooldown, and 40 minutes of functional, self-paced exercises. In the video, 2 healthcare professionals demonstrate a lower and higher difficulty level of each exercise. The program starts with a level 1 video and switches to a level 2 video midway.
  A registered healthcare professional, called the healthcare partner, visits select classes and serves as a resource to participants and facilitators.
  Arms: TIME at Home

SUMMARY:
The goal of this randomized controlled trial is to compare the short-term effects of a virtual, community-based, task-oriented group exercise program (TIME™ at Home) with a waitlist control in community-dwelling adults with balance and mobility limitations.

The main questions the trial aims to answer are:

1. Will there be improvements in physical and mental health outcomes, and caregiver mood and assistance, following participation in the TIME™ at Home exercise program that are greater than in the waitlist control group?
2. Will level of mobility limitation, sex, or gender influence the experiences of people in the exercise program?
3. What will be the costs of the TIME™ at Home exercise program for the organization delivering the program, and the people who are in the exercise program?

Participants and their caregivers will be asked to complete 3 evaluations using Zoom at study entry and 2 and 5 months later.

* Participants will complete tests of balance and walking and questionnaires.
* Caregivers will only complete questionnaires.

After the first evaluation, participants will be randomly assigned to either participate in:

* the 8-week TIME™ at Home exercise program from their homes using Zoom, or
* to wait 5 months (waitlist control group) before beginning the 8-week TIME™ at Home exercise program

DETAILED DESCRIPTION:
Mobility limitations are highly prevalent, limit everyday functioning, and increase the need for caregiver assistance in people with chronic health conditions, such as stroke, and multiple sclerosis. While community exercise programs have been shown to improve physical and mental health, older adults with mobility limitations face numerous challenges with attending in-person community exercise programs. Challenges relate to the availability and cost of transportation, inclement weather, inadequate building access, program cost, risk of infection, and pandemic-related program closures. In addition, caregivers commonly need to provide transportation, which can take time away from paid employment and other daily activities. Some recreation centres do not have the funding to operate exercise programs for people with balance and mobility limitations that require instructors with specialized skills and a high level of exercise supervision.

The objectives of the TIME™ at Home randomized controlled trial are:

1. To estimate the short-term effects of a virtual, community-based, task-oriented group exercise program (TIME™ at Home) compared to a waitlist control on improving everyday function (primary outcome), mobility, well-being, reliance on walking aids, caregiver assistance, caregiver mood, and caregiver confidence in care-recipient balance (secondary outcomes) in community-dwelling adults with mobility limitations;
2. To determine whether level of mobility limitation, sex, or gender, modifies the effect of the TIME™ at Home program compared to a waitlist control in improving everyday function;
3. To assess the cost-effectiveness of the TIME™ at Home program from a societal perspective; and
4. To explore exercise participants', caregivers' and program providers' experiences during the intervention phase.

ELIGIBILITY:
Inclusion Criteria:

1. adult defined as age 18 years or older;
2. mobility limitations (eg, need to use a walking aid, difficulty stepping onto curbs, ramps, stairs, or walk on uneven surfaces);
3. living independently in the community (in own home or assisted living settings);
4. able to walk a minimum of 10 metres independently (with walking aids if used) without assistance and/or supervision from another person;
5. able to stand up from and sit down onto a chair independently, without supervision;
6. able to maintain balance while exercising in standing (e.g., marching on the spot) holding onto the back of a chair or a sturdy countertop;
7. has a study partner (e.g., caregiver, family member or friend) willing to be present, at minimum, during the first evaluation in the home via Zoom;
8. able to speak and read English to understand informed consent and follow instructions for study procedures and exercises;

Exclusion Criteria:

1. involvement in another formal exercise or rehabilitation program in the next 2 months;
2. previous participation in the TIME at Home exercise program;
3. health conditions or symptoms preventing participation in exercise;
4. cognitive impairment, defined as a score of <11/15 on the 5-minute Montreal Cognitive Assessment (MoCA);
5. severe visual impairment;
6. severe hearing impairment

Caregivers

Inclusion criteria:

1. caregiver defined as an individual who helps the exercise participant to live at home by providing support and assistance with at least one basic (e.g., self-care) and/or instrumental activity of daily living (e.g., doing groceries, cleaning, managing finances, making meals, doing laundry, etc.) at least once a week;
2. able to speak and read English.

Exclusion criteria:

1. Is a paid personal support worker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Subjective Index of Physical and Social Outcome-Physical scale (SIPSO-P) from baseline to 2 months | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Score from 0 to 20 points, 5-item self-report scale measuring everyday functioning

SECONDARY OUTCOMES:
7-item Berg balance scale (7BBS) | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Score from 0 to 28 points on 7-item performance-based measure
30-second sit-to-stand test (30STS) | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Number of stands completed in 30 seconds
Timed 'up and go' (TUG) test | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Time in seconds, taken to stand up from a standard armchair, walk a distance of 3 metres, turn around, walk back to the chair, and sit down again
3-metre walk test (3mWT, comfortable pace) | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Comfortable walking speed in metres/second based on time taken to walk 3 metres
3-metre walk test (3mWT, fast pace) | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Fast walking speed in metres/second based on time taken to walk 3 metres
2-minute step test (2ST) | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Number of times the knee reaches the required height in 2 minutes
Activities-specific balance confidence (ABC) scale | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Score from 0 to 100 points on the 16-item self-report scale
Center for epidemiological studies depression (CES-D) scale | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Score from 0 to 60 points on the 20-item self-report scale
PROMIS v2.0 Social Isolation short form | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Score from 0 to 20 points on the 4-item self-report scale
EuroQoL-5D-5L visual analog scale (EQ-VAS) | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Score from 0 to 100 points on the visual analog scale
Caregiver Assistance Scale (CAS) | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Score from 0 to 102 points on the 17-item self-report scale, completed by caregiver
Center for epidemiological studies depression (CES-D) scale-Caregiver | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Score from 0 to 60 points on the 20-item self-report scale, completed by caregiver
Activities-specific balance confidence (ABC) scale-Caregiver | 0 months (baseline), 2 months (immediately post-intervention), and 5 months (3 months post-intervention)
  Score from 0 to 100 points on the 16-item self-report scale, completed by caregiver
Program delivery cost | 2 months (immediately post-intervention)
  Cost ($) for community organizations to run the TIME at Home program in the Experimental group
Cost ($) of exercise participation | 2 months (immediately post-intervention)
  Cost ($) for a participant in the Experimental group to participate in the TIME at Home program
Amount ($) willing to pay to register for TIME at Home | 2 months (immediately post-intervention)
  Amount ($) that participants in the Experimental group would be willing to pay out-of-pocket to receive the program
Quality-adjusted life-years (QALYs) | 2 months (immediately post-intervention)
  Scores on the EQ-5D-5L convert to a single index value used to calculate quality-adjusted life-years (QALYs)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Salbach, PhD, Principal Investigator — University of Toronto
Locations (4):
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - Bruyère Research Institute, Ottawa, Ontario
  - University of Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
The anonymized data collected during the study, the trial protocol, statistical analysis plan, and informed consent form, will be shared with qualified researchers engaging in REB-approved independent scientific research, upon request to the research team.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study ends.
Access Criteria: Please contact the research team

REFERENCES:
- [Derived] Salbach NM, Jones CA, Barclay R, Sveistrup H, Sheehy L, Bayley MT, Inness EL, Legasto-Mulvale JM, Barbosa Dos Santos R, Fung J, Moineddin R, Teasell RW, Catizzone M, Hovanec N, Cameron JI, Munce S, O'Neil J, Jaglal SB, Aravind G, Su TT, Hanson HM. Short-term effects of a virtual, community-based, task-oriented group exercise programme incorporating a healthcare-community partnership compared to a waitlist control on increasing everyday function among adults with mobility limitations: protocol for the TIME at Home randomised controlled trial. BMJ Open. 2025 Jul 28;15(7):e102694. doi: 10.1136/bmjopen-2025-102694. PMID 40721264